CLINICAL TRIAL: NCT07305155
Title: A Feasibility Randomized-controlled Trial Comparing Trauma-focused Mentalization Based Treatment With Standard Mentalization-based Treatment in Patients Presenting With Complex Post-traumatic Stress and Borderline Personality Disorder
Brief Title: Pilot Study for the Evaluation of a New Psychotherapeutic Treatment for Borderline Personality Disorder Patients With Post-traumatic Stress Symptoms
Acronym: MBT-TF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eva Rüfenacht (Other)
Responsible Party: Sponsor-Investigator, Eva Rüfenacht, Senior Physician, Head of the Emotion Regulation Disorders Unit , Principal Investigator, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025-01307
Record Dates: First submitted 2025-11-28; First posted 2025-12-26 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Borderline Personality Disorder (BPD); PTSD - Post Traumatic Stress Disorder
Keywords: Borderline Personality Disorder; Post Traumatic Stress Disorder; Mentalization-based treatment; trauma-focused mentalization-based treatment
MeSH Terms: conditions — Borderline Personality Disorder; Combat Disorders; Stress Disorders, Post-Traumatic | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This study is a monocentric, two-arm feasibility randomised controlled trial (RCT), comparing the intervention (MBT-TF) with TAU (standard MBT).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stardard Mentalization-Based Treatment (Active Comparator)
  Interventions: Other: Standard Mentalization-Based Treatment
- Trauma-Focused Mentalization-Based Treatment (Experimental)
  Interventions: Other: Trauma-Focused Mentalization-Based Treatment

INTERVENTIONS:
Other: Standard Mentalization-Based Treatment — Standard MBT treatment, specialized and validated treatment for BPD, which consists of weekly group and individual sessions for one year without any trauma focus, will serve as a comparison.
  Other Names: TAU (Treatment As Usual); Standard MBT
  Arms: Stardard Mentalization-Based Treatment
Other: Trauma-Focused Mentalization-Based Treatment — The intervention will be a trauma-focused Mentalization-based treatment (MBT-TF), consisting of a 3-phase group intervention with an individual component (weekly sessions) offered as needed, focused psychoeducation about post-traumatic stress symptoms and on improving trauma related mentalizing abilities and interpersonal functioning over a 12-month period (45-50 sessions in total).
  Arms: Trauma-Focused Mentalization-Based Treatment

SUMMARY:
Borderline Personality Disorder (BPD) is a serious mental health condition that often co-occurs with Complex PTSD (CPTSD), making treatment more challenging. Trauma-Focused Mentalization-Based Treatment (MBT-TF) is a new adaptation of standard MBT designed for individuals with high trauma exposure. Early findings are promising, but further research is needed. This study at Geneva University Hospitals (HUG) will test the feasibility and acceptability of MBT-TF compared with standard MBT, gathering feedback from patients and clinicians and laying the groundwork for a larger clinical trial.

DETAILED DESCRIPTION:
Borderline Personality Disorder (BPD) is a serious mental health condition that can make it difficult for people to regulate emotions and maintain relationships. Even with specialised therapy, many individuals with BPD continue to experience significant difficulties in daily life.

A large proportion of patients with BPD also show symptoms of trauma, such as Post-Traumatic Stress Disorder (PTSD) or its more complex form (CPTSD). About half of all patients with BPD meet the criteria for CPTSD, and this overlap may partly explain why standard treatments are sometimes less effective. At present, there are no clear treatment guidelines for people who have both BPD and CPTSD, even though this combination greatly affects quality of life and social functioning.

Mentalization-Based Treatment (MBT) is a structured therapy developed in the 1990s for BPD. A newer version, Trauma-Focused MBT (MBT-TF), has been designed for individuals with high levels of trauma or CPTSD. Early results from MBT-TF are promising, but further research is needed before a large-scale trial can be undertaken.

This upcoming study at Geneva University Hospitals (HUG) will examine whether MBT-TF can be delivered effectively and accepted by both patients and clinicians, compared with standard MBT ("treatment as usual"). It will also gather early evidence on whether MBT-TF may be more effective. An independent steering committee of international experts and a patient representative will oversee the trial.

Patients will be followed during 15 months, including 1 year of treatment. Patients will have to fill in questionnaires, and follow individual interviews. In total, 5 visits will be performed for the study, in addition to the stardard clinical follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years.
* Meeting ≥4 of 9 SCID-5 PD criteria associated with functional impairment (either subthreshold or full BPD diagnosis), and an LPFS-BF 2.0 score ≥31 (≥1.5 standard deviations above the latent mean, T-score ≥65), indicating moderate to severe personality disorder features.
* Diagnosis of CPTSD according to ICD-11 criteria, confirmed via ITQ with clinical checks.

Exclusion Criteria:

* Mental disability.
* Severe psychiatric psychopathology requiring immediate treatment (e.g., BMI <16.5, acute bipolar episode, current psychosis).
* Severe active substance dependence.
* Severe physical health problems (e.g., severe cardiovascular conditions). Severe neurological disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2030-09-01 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | Through study completion, an average of 3 years
  Proportion of recruited eligible patients

SECONDARY OUTCOMES:
Non-eligibility rate | Through study completion, an average of 3 years
  proportion of eligible patients not included
Proportion of included but untreated patients | Through study completion, an average of 3 years
  Screening failures
Mean pre-treatment and 15-month follow-up differences in CAPS-5 or ITQ CPTSD with clinical checks scores | Baseline and 15 months post-randomisation
Proportion of patients initiating MBT-TF within three months of recruitment | Through study completion, an average of 3 years
Number of days between randomisation and first MBT-TF session | Randomization and First Treatment Day
Proportion of missing or incomplete questionnaire responses assessing psychological and social aspects | Through study completion, an average of 3 years
Proportion of losses to follow-up | Through study completion, an average of 3 years
Treatment completion rate | Through study completion, an average of 3 years
  Rate of patients completing 8 months of treatment
Mean number of sessions attended | Through study completion, an average of 3 years
Patient expectation and credibility score | At baseline and at 15 months post randomisation
  Patient expectation and credibility assessed with validated scale ("The French credibility/expectancy questionnaire"). This questionnaire has a two-factor structure, and includes six items assessing credibility (3) and expectancy (3), with a higher score indicating higher credibility and/or expectancy.
Patient satisfaction score | 15 months post-randomization
  Patient satisfaction score is assessed with the validated "Client Satisfaction Questionnaire (CSQ-8)"). The questionnaire evaluates client satisfaction based on 8 questions and on a 4-point Lickert scale (1 = unsatisfied, 4 = satisfied). Higher score indicates higher satisfaction.
Frequency of serious adverse events | Baseline, 9 months, 15 months, 18 months post randomisation
Average therapist adherence scores across sessions for both arms using a standardised adherence scale | 15 months post-randomisation
  Therapist fidelity to MBT-TF and standard MBT will be assessed using the French version of the MBT-Adherence and Competence Scale (MBT-ACS) and a complementary MBT-TF-specific rating. The average therapist adherence scores will be assessed across sessions for both arms (0-5, "0 = no adherence", "5 = full adherence") measuring fidelity to key protocol components, including therapeutic techniques, session structure, and mentalizing interventions.
Mean change in CAPS-5 total score | At baseline and at 15 months post-randomisation
  Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Rating ranges from 0 (absent) to 4 (extreme/incapacitating) for each of the 20 items. Total symptom severity score is calculated by summing scores for all items.
Mean change in ITQ CPTSD with clinical checks total symptom score | At baseline and at 15 months post-randomisation
  ITQ: International Trauma Questionnaire with clinical checks Scoring based on a 0-4 Likert scale ('Not at all' to 'Extremely') for each item (18 in total), higher scores indicating greater severity

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Geneva, Geneva, Canton of Geneva, Switzerland